CLINICAL TRIAL: NCT01542632
Title: A Randomized, Phase 1b Study to Investigate the Safety and Immunogenicity of Various Schedules of Tetravalent Chimeric Dengue Vaccine in Healthy Adult Volunteers Between the Ages of 18 - 45 Years
Brief Title: A Comparison of the Safety and Immunogenicity of Various Schedules of Dengue Vaccine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INV-DEN-104; U1111-1177-8166 (Registry Identifier: WHO)
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: safety and immunogenicity of dengue vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): Takeda's Tetravalent Dengue Vaccine Candidate (TDV), 0.5 mL, subcutaneous injection in one arm and placebo, 0.5 mL, subcutaneous injection in the other arm on Day 0. TDV, 0.5 mL, subcutaneous injection on Day 90.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV); Drug: Placebo
- Group 2 (Experimental): TDV, 0.5 mL, subcutaneous injection in one arm and TDV 0.5 mL, subcutaneous injection in the other arm on Day 0. Placebo, 0.5 mL, subcutaneous injection on Day 90.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV); Drug: Placebo
- Group 3 (Experimental): TDV, 0.5 mL, subcutaneous injection in one arm and TDV, 0.5 mL, subcutaneous injection in the other arm on Day 0. TDV, 0.5 mL, subcutaneous injection on Day 90.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV)
- Group 4 (Experimental): TDV new formulation, 0.5 mL, subcutaneous injection in one arm and new formulation placebo, 0.5 mL, subcutaneous injection in the other arm on Days 0 and 90.
  Interventions: Biological: TDV New Formulation; Drug: New Formulation Placebo
- Group 5 (Experimental): TDV new formulation, 0.5 mL, subcutaneous injection in one arm and TDV new formulation, 0.5 mL, subcutaneous injection in the other arm on Days 0 and 90.
  Interventions: Biological: TDV New Formulation; Drug: New Formulation Placebo
- Group 6 (Experimental): 1/10 TDV, 0.5 mL, subcutaneous injection on Days 1 and 90.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV)

INTERVENTIONS:
Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV) — TDV subcutaneous injection
  Arms: Group 1; Group 2; Group 3; Group 6
Biological: TDV New Formulation — TDV New Formulation subcutaneous injection
  Arms: Group 4; Group 5
Drug: Placebo — Placebo subcutaneous injection
  Arms: Group 1; Group 2
Drug: New Formulation Placebo — New Formulation placebo subcutaneous injection
  Arms: Group 4; Group 5

SUMMARY:
A Phase 1 study to compare the safety, tolerability and immunogenicity of different dose schedules of subcutaneously (SC) administered dengue vaccine in healthy adults and to compare the immunogenicity of different dose schedules of the vaccine.

Blood samples were obtained for safety labs on Days 0, 7, 14, 90, 97, 104 and measurement of viremia at baseline [during the screening period or on day of vaccination (Day 0)], and then on Days 7, 9, 11, 14, 17, 21, 90, 97, and 104. Blood samples for measurement of dengue neutralizing antibodies in serum were obtained at baseline [during the screening period or on day of vaccination (Day 0)], then on Days 30, 90 and 120.

The entire duration for each individual subjects participation was approximately 5 months including recruitment and collection of data for primary outcomes (through Day 120).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years and ≤ 45 years old at time of screening
2. In good health as determined by medical history, physical examination including height and weight
3. Normal clinical safety laboratory examinations [Sodium (Na), Potassium (K), Glucose, Blood Urea Nitrogen (BUN), creatinine, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), total bilirubin, White Blood Cell (WBC), neutrophil count, hemoglobin, platelets, Prothrombin Time (PT), Partial Thromboplastin Time (PTT), and urinalysis (by dipstick)].
4. Weight: Body Mass Index (BMI) ≤32
5. Blood tests negative for antibodies to Human Immuno-virus (HIV-1), Hepatitis C, and Hepatitis B surface antigen

Exclusion Criteria:

1. Any condition which would limit the subject's ability to complete the study in the opinion of the Investigator
2. Clinically significant ECG findings
3. History of any significant dermatologic disease in the last 6 months,
4. History of diabetes mellitus
5. History of recurring headaches or migraines (more frequent than once per week) or on prescription medication for treatment of recurring headaches or migraines
6. Hypersensitivity to any vaccine
7. Receipt of any vaccine in the 4 weeks preceding the first vaccination
8. Planned receipt of any vaccine in the 4 weeks following each of the vaccinations in this study
9. Known history of Japanese Encephalitis Virus (JEV) and/or Yellow Fever (YF)
10. Previous vaccination (in a clinical trial or with an approved product) against flaviviruses including dengue, yellow fever (YF) and Japanese Encephalitis (JE)
11. Seropositivity to dengue or West Nile (WN) virus
12. Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months
13. Use within the previous 6 months of systemic corticosteroids therapy (at a dose of at least 0.5 mg/kg/day). Topical prednisone is not permitted if currently in use or within the last 3 months. Note, inhaled prednisone (or equivalent) is allowed
14. Use of any non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen or antihistamines for the 3 days immediately prior to each vaccination
15. Use of any prescription or over the counter medications (besides those specifically mentioned above or those required for medical management of concurrent diseases) 7 days before the first vaccination (Day 0)
16. Positive urine screen for cocaine, amphetamines, opiates, or cannabinoids
17. Donation of blood 6 weeks before the first dose(s) (Day 0) until 30 days after the dose on day 90
18. Females who are pregnant or lactating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2014-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Gordon, MD, Study Director — Inviragen Inc.
Locations (3):
- United States (3):
  - Heart Center of the Rockies, Fort Collins, Colorado
  - University of Texas Medical Branch, Galveston, Texas
  - Advanced Clinical Research, West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 23 January 2012 to 10 January 2014.
Pre-assignment Details: Participants were enrolled in 1 of 6 treatment groups (GRP). GRP1: 1 dose TDV on Day 0 and 90, GRP2: 2 doses of TDV on Day 0, GRP3: 2 Doses of TDV on Day 0 and 1 dose of TDV on Day 90, GRP4: 1 Dose of TDV New Formula on Day 0 and 90, GRP5: 2 doses of TDV New Formula on Day 0 and 90 and GRP6: 1/10 dose of TDV on Day 0 and 90.
Groups:
- Group 1 (D0:TDV,P D90:TDV): Takeda's Tetravalent Dengue Vaccine Candidate (TDV), 0.5 mL, subcutaneous injection in one arm and TDV placebo (P), 0.5 mL, subcutaneous injection in the other arm on Day 0 (D0). TDV, 0.5 mL, subcutaneous injection on Day 90 (D90).
- Group 2 (D0:TDV,TDV D90:P): TDV, 0.5 mL, subcutaneous injection in one arm and TDV, 0.5 mL, subcutaneous injection in the other arm on Day 0. TDV placebo, 0.5 mL, subcutaneous injection on Day 90.
- Group 3 (D0:TDV,TDV D90:TDV): TDV, 0.5 mL, subcutaneous injection in one arm and TDV, 0.5 mL, subcutaneous injection in the other arm on Day 0. TDV, 0.5 mL, subcutaneous injection on Day 90.
- Group 4 (D0:TDVN,P D90:TDVN,P): TDV new formulation(TDVN), 0.5 mL, subcutaneous injection in one arm and TDV new formulation placebo, 0.5 mL, subcutaneous injection in the other arm on Days 0 and 90.
- Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN): TDV new formulation, 0.5 mL, subcutaneous injection in one arm and TDV new formulation, 0.5 mL, subcutaneous injection in the other arm on Days 0 and 90.
- Group 6 (D0:1/10TDV D90:1/10TDV): 1/10 TDV, 0.5 mL, subcutaneous injection on Days 0 and 90.
Period: Overall Study
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV)
Started | 25 | 25 | 24 | 21 | 21 | 24
Completed | 25 | 24 | 23 | 19 | 17 | 24
Not Completed | 0 | 1 | 1 | 2 | 4 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 2 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor/Investigator Decision | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 2 (DO:TDV,TDV D90:P): TDV, 0.5 mL, subcutaneous injection in one arm and TDV, 0.5 mL, subcutaneous injection in the other arm on Day 0. TDV placebo, 0.5 mL, subcutaneous injection on Day 90.
- Total: Total of all reporting groups
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (DO:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV) | Total
Number analyzed (Participants) | 25 | 25 | 24 | 21 | 21 | 24 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (5.74) | 28.2 (6.36) | 29.2 (6.40) | 30.0 (6.67) | 30.3 (7.95) | 32.5 (6.04) | 30.0 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 12 | 8 | 9 | 9 | 67
  Male | 10 | 11 | 12 | 13 | 12 | 15 | 73
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Black/African American | 0 | 2 | 1 | 0 | 0 | 1 | 4
  Hawaiian/Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hispanic Or Latino | 6 | 3 | 7 | 0 | 2 | 0 | 18
  Other | 2 | 0 | 1 | 0 | 0 | 0 | 3
  White | 17 | 19 | 14 | 20 | 19 | 23 | 112
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 24 | 21 | 21 | 24 | 140
Weight [Mean (Standard Deviation); unit: kg] | 73.3 (11.66) | 75.9 (13.22) | 76.7 (15.76) | 80.8 (14.12) | 77.3 (14.91) | 81.7 (16.02) | 77.5 (14.36)
Height [Mean (Standard Deviation); unit: m] | 1.71 (0.092) | 1.71 (0.084) | 1.70 (0.108) | 1.76 (0.105) | 1.73 (0.099) | 1.75 (0.104) | 1.72 (0.100)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.81 (2.423) | 25.97 (3.314) | 26.50 (3.735) | 26.09 (3.202) | 25.81 (3.712) | 26.35 (3.517) | 25.91 (3.323)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Injection Site Reactions Following Either Vaccine Dose Worst Severity Reported
Description: Erythema and Edema Were Graded Per The FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Where Grade 0=none to Grade 4=Severe. Pain and Itching were graded using Common Terminology Criteria for Adverse Events (CTCAE) 4.03 where Grade 0=no pain or itching to Grade 4= Life-threatening/severe. Only those score categories for which there was at least 1 participant are reported.
Time Frame: Day 0 to Day 104
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Group 3 (D0:TDV,TDV D90:TDV): TDV, 0.5 mL, subcutaneous injection in one arm and TDV, 0.5 mL, subcutaneous injection in the other arm on Day 1. TDV, 0.5 mL, subcutaneous injection on Day 90.
- Group 4 (D0:TDVN,P D90:TDVN,P): TDV new formulation (TDVN), 0.5 mL, subcutaneous injection in one arm and TDV new formulation placebo, 0.5 mL, subcutaneous injection in the other arm on Days 0 and 90.
- Group 6 (D0:1/10TDV D90:1/10TDV): 1/10 TDV, 0.5 mL, subcutaneous injection on Days 1 and 90.
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV)
Number analyzed (Participants) | 25 | 25 | 24 | 21 | 21 | 24
participants
  Edema=0 | 25 | 25 | 24 | 21 | 21 | 24
  Erythema=0 | 25 | 25 | 24 | 21 | 21 | 24
  Itching=0 | 24 | 19 | 23 | 20 | 21 | 22
  Itching=1 | 1 | 6 | 1 | 1 | 0 | 2
  Pain=0 | 19 | 18 | 19 | 16 | 18 | 20
  Pain=1 | 6 | 7 | 4 | 5 | 2 | 4
  Pain=2 | 0 | 0 | 1 | 0 | 1 | 0

2. Secondary Outcome: Percentage of Participants With Serotype-Specific TDV Viral RNA Detected After First and Second Vaccinations
Description: Serotype-Specific TDV Viral RNA was assessed for the four dengue serotypes: Dengue-1, Dengue-2, Dengue-3 and Dengue-4 . Only those serotypes and time-points where at least 1 participant had Serotype-Specific TDV Viral RNA Detected is reported.
Time Frame: various timepoints up to 30 days after each dose (Up to Day 120)
Population: Full Analysis Set included all enrolled participants.
Measure: Number; unit: percentage of participants
Groups:
- Group 1 (D0:TDV,P D90:TDV): Takedas Tetravalent Dengue Vaccine Candidate (TDV), 0.5 mL, subcutaneous injection in one arm and TDV placebo (P), 0.5 mL, subcutaneous injection in the other arm on Day 0 (D0). TDV, 0.5 mL, subcutaneous injection on Day 90 (D90).
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV)
Number analyzed (Participants) | 25 | 25 | 24 | 21 | 21 | 24
percentage of participants
  Day 7 Dengue-2 | 20 | 8 | 12 | 19 | 19 | 16
  Day 9 Dengue-2 | 56 | 72 | 66 | 47 | 61 | 45
  Day 9 Dengue-3 | 0 | 0 | 0 | 4 | 0 | 0
  Day 11 Dengue-2 | 64 | 68 | 75 | 61 | 52 | 70
  Day 11 Dengue-3 | 0 | 0 | 0 | 4 | 0 | 0
  Day 11 Dengue-4 | 0 | 0 | 0 | 4 | 0 | 0
  Day 14 Dengue-2 | 52 | 52 | 66 | 33 | 28 | 41
  Day 17 Dengue-1 | 0 | 0 | 0 | 4 | 0 | 0
  Day 17 Dengue-2 | 24 | 12 | 8 | 14 | 0 | 12
  Day 21 Dengue-2 | 0 | 0 | 0 | 4 | 0 | 0
  Day 90 Dengue-3 | 0 | 4 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With at Least 1 Adverse Event Following Either Vaccine Dose
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
Time Frame: For 30 days after each dose (Up to Day 120)
Population: Safety Population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV)
Number analyzed (Participants) | 25 | 25 | 24 | 21 | 21 | 24
participants | 22 | 19 | 21 | 17 | 17 | 18

4. Primary Outcome: Number of Participants With at Least 1 Adverse Events Related to TDV Following Either Vaccine Dose
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. Some AEs are automatically considered related because of temporal relationship to vaccination.
Time Frame: For 30 days after each dose (Up to Day 120)
Population: Safety Population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV)
Number analyzed (Participants) | 25 | 25 | 24 | 21 | 21 | 24
participants | 20 | 16 | 18 | 14 | 12 | 14

5. Secondary Outcome: Geometric Mean Neutralizing Antibody Titers (GMTs) of All Four Dengue Serotypes
Time Frame: Days 30, 90 and 120 after 1st vaccination
Population: Participants from the Full Analysis, all enrolled participants, with data available for analysis at the given time-point.
Measure: Geometric Mean (Standard Deviation); unit: titer
Groups:
- Group 4 (D0:TDV,P D90:TDV,P): TDV new formulation (TDVN), 0.5 mL, subcutaneous injection in one arm and TDV new formulation placebo, 0.5 mL, subcutaneous injection in the other arm on Days 0 and 90.
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDV,P D90:TDV,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV)
Number analyzed (Participants) | 25 | 25 | 24 | 21 | 21 | 24
titer
  Day 30 Dengue-1 (n=25, 24, 24, 21, 19, 24) | 428.6 (2.28) | 473.6 (2.60) | 370.1 (3.87) | 45.6 (3.97) | 69.1 (5.51) | 391.4 (3.30)
  Day 30 Dengue-2 (n=25, 24, 24, 21, 19, 24) | 6411.9 (7.83) | 4843.3 (3.42) | 6274.1 (3.57) | 4953.8 (3.01) | 5419.6 (3.06) | 7315.3 (5.90)
  Day 30 Dengue-3 (n=25, 24, 24, 21, 19, 24) | 62.3 (5.78) | 151.0 (4.12) | 70.3 (6.10) | 47.2 (5.69) | 62.0 (6.19) | 37.4 (6.13)
  Day 30 Dengue-4 (n=25, 24, 24, 21, 19, 24) | 8.2 (2.20) | 19.4 (4.65) | 11.6 (5.00) | 45.6 (5.13) | 21.5 (5.89) | 17.4 (10.28)
  Day 90 Dengue-1 (n=25, 24, 23, 20, 18, 23) | 155.6 (4.26) | 130.7 (2.75) | 142.2 (6.16) | 27.3 (3.11) | 37.0 (5.91) | 127.6 (5.92)
  Day 90 Dengue-2 (n=25, 24, 23, 20, 18, 23) | 1597.9 (2.81) | 1758.7 (3.29) | 1814.4 (3.13) | 1383.1 (2.82) | 1288.7 (3.14) | 1756.5 (5.80)
  Day 90 Dengue-3 (n=25, 24, 23, 20, 18, 23) | 32.0 (4.10) | 44.9 (4.04) | 28.7 (5.38) | 20.0 (4.17) | 27.7 (4.68) | 22.6 (4.87)
  Day 90 Dengue-4 (n=25, 24, 23, 20, 18, 23) | 6.6 (1.76) | 10.3 (3.44) | 9.4 (3.62) | 13.7 (3.60) | 11.2 (3.62) | 13.5 (6.85)
  Day 120 Dengue-1 (n=25, 24, 23, 19, 17, 24) | 223.2 (3.55) | 136.5 (3.88) | 216.3 (6.23) | 38.6 (2.70) | 65.4 (5.00) | 179.6 (4.85)
  Day 120 Dengue-2 (n=25, 24, 23, 19, 17, 24) | 1597.9 (2.27) | 1478.9 (2.72) | 1893.9 (2.89) | 1631.8 (3.49) | 1295.5 (3.22) | 1356.1 (5.37)
  Day 120 Dengue-3 (n=25, 24, 23, 19, 17, 24) | 51.3 (2.28) | 42.4 (3.70) | 56.6 (4.43) | 30.5 (3.36) | 51.2 (3.00) | 25.9 (3.87)
  Day 120 Dengue-4 (n=25, 24, 23, 19, 17, 24) | 11.5 (2.50) | 8.9 (2.70) | 12.0 (3.58) | 23.2 (3.52) | 25.5 (3.74) | 12.8 (5.81)

6. Primary Outcome: Rate of Seroconversion to Each of Four Dengue Serotypes
Description: Rate of seroconversion was defined as the percentage of participants with Plaque Reduction Neutralization Test titer resulting in 50 % reduction in Plagues (PRNT50) titer ≥ 10 for participants seronegative at Baseline or a greater than four-fold increase in PRNT50 for participants seropositive at Baseline.
Time Frame: Up to 30 days after the last immunization (Up to Day 120)
Population: Participants from the Full Analysis Set, all enrolled participants, with data available at the given time-point.
Measure: Number; unit: percentage of participants
Groups:
- Group 6 (D0:1/10TDV D90:1/10TDV: 1/10 TDV, 0.5 mL, subcutaneous injection on Days 0 and 90.
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV
Number analyzed (Participants) | 25 | 25 | 24 | 21 | 19 | 24
percentage of participants
  Dengue-1 Day 30 (n=25, 24, 24, 21, 19, 24) | 100.0 | 95.8 | 100.0 | 81.0 | 89.5 | 100.0
  Dengue-2 Day 30 (n=25, 24, 24, 21, 19, 24) | 96.0 | 100.0 | 100.0 | 100.0 | 100.0 | 95.8
  Dengue-3 Day 30 (n=25, 24, 24, 21, 19, 24) | 84.0 | 100.0 | 87.5 | 85.7 | 94.7 | 66.7
  Dengue-4 Day 30 (n=25, 24, 24, 21, 19, 24) | 36.0 | 58.3 | 33.3 | 81.0 | 57.9 | 29.2
  Dengue-1 Day 90 (n=25, 24, 23, 20, 18, 24) | 96.0 | 91.7 | 95.7 | 75.0 | 72.2 | 87.5
  Dengue-2 Day 90 (n=25, 24, 23, 20, 18, 24) | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 91.7
  Dengue-3 Day 90 (n=25, 24, 23, 20, 18, 24) | 80.0 | 91.7 | 82.6 | 75.0 | 83.3 | 62.5
  Dengue-4 Day 90 (n=25, 24, 23, 20, 18, 24) | 24.0 | 29.2 | 21.7 | 50.0 | 38.9 | 37.5
  Dengue-1 Day 120 (n=25, 24, 23, 19, 17, 24) | 100.0 | 95.8 | 95.7 | 84.2 | 94.1 | 95.8
  Dengue-2 Day 120 (n=25, 24, 23, 19, 17, 24) | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 95.8
  Dengue-3 Day 120 (n=25, 24, 23, 19, 17, 24) | 100.0 | 95.8 | 91.3 | 94.7 | 94.1 | 83.3
  Dengue-4 Day 120 (n=25, 24, 23, 19, 17, 24) | 60.0 | 33.3 | 52.2 | 73.7 | 76.5 | 41.7

ADVERSE EVENTS:
Time Frame: Day 0 to Day 120
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Group 1 (D0:TDV,P D90:TDV) | Group 2 (D0:TDV,TDV D90:P) | Group 3 (D0:TDV,TDV D90:TDV) | Group 4 (D0:TDVN,P D90:TDVN,P) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) | Group 6 (D0:1/10TDV D90:1/10TDV)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/21 | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 24/25 | 18/25 | 20/24 | 16/21 | 17/21 | 18/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (D0:TDV,P D90:TDV) (N=25) | Group 2 (D0:TDV,TDV D90:P) (N=25) | Group 3 (D0:TDV,TDV D90:TDV) (N=24) | Group 4 (D0:TDVN,P D90:TDVN,P) (N=21) | Group 5 (D0:TDVN,TDVN D90:TDVN,TDVN) (N=21) | Group 6 (D0:1/10TDV D90:1/10TDV) (N=24)
Fatigue (General disorders) | 13 | 11 | 9 | 10 | 10 | 7
Injection site haematoma (General disorders) | 1 | 2 | 4 | 0 | 0 | 0
Pain (General disorders) | 0 | 3 | 2 | 1 | 0 | 1
Headache (Nervous system disorders) | 14 | 13 | 12 | 10 | 12 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 8 | 4 | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5 | 1 | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 0 | 0 | 5 | 6 | 6
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 6 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 2 | 3 | 4 | 2
Eye pain (Eye disorders) | 2 | 3 | 2 | 5 | 4 | 4
Photophobia (Eye disorders) | 2 | 3 | 2 | 3 | 5 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 2 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.